CLINICAL TRIAL: NCT06594497
Title: The Effect of Motor Imagery Training on Knee Functions and Kinesiophobia in Football Players With Anterior Cruciate Ligament Repair
Brief Title: Motor Imagery Training Football Players With Anterior Cruciate Ligament Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/09-34
Record Dates: First submitted 2024-07-31; First posted 2024-09-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-07

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physiotherapy group (Active Comparator): In line with the relevant physician's protocol, Quadriceps Isometric Exercises, Passive ROM exercises, active hip exercises while wearing a brace, ankle exercises, and ice application training are given. The patient is asked to continue as a home program for 2 weeks. After 2 weeks, electrical stimulation (15-20 minutes), current exercises, and ice application continue in the unit. (15min). A total of 30 sessions are applied. In addition, it is requested that the exercises be done at home, as in the treatment program (3x10).
  Interventions: Other: Conventional Physiotherapy
- Conventional Physiotherapy + Kinesthetic motor imagery training group (Experimental): Motor imagery training will be planned according to the PETTLEP model. A quiet environment will be provided to minimize distractions during the motor imagery session, and the patient's eyes will be closed throughout the session. At the very beginning of the session, a relaxation exercise lasting approximately 2 minutes will be performed to maximize attention during motor imagery. In relaxation exercises, patients will be asked to focus on their breathing, become aware of each body area, and relax the muscles in these areas. Care will be taken to ensure that the imagined movement is of similar duration to the real and optimal movement. Motor imagery will mostly be studied from a first-person perspective. During kinesthetic imagery, people will be asked to feel the movement of their body parts during each exercise without any body movement occurring. 3 sessions per week will last for 6 weeks in total.
  Interventions: Other: Conventional Physiotherapy; Other: Conventional Physiotherapy + Kinesthetic motor imagery training

INTERVENTIONS:
Other: Conventional Physiotherapy — Conventional Physiotherapy
Other: Conventional Physiotherapy + Kinesthetic motor imagery training — Conventional Physiotherapy + Kinesthetic motor imagery training
  Arms: Conventional Physiotherapy + Kinesthetic motor imagery training group

SUMMARY:
Volunteer participants who have undergone anterior cruciate ligament surgery at Bursa Çekirge State Hospital and meet the inclusion criteria will be included in the study. The study will select a sample group from the universe using the probability sampling method (simple random sampling). Participants will be divided into 2 groups: Conventional Physiotherapy + Kinesthetic motor imagery training group and Conventional physiotherapy group with randomization software (https://www.randomizer.org/). Conventional physiotherapy practices created by the physician will be applied by physiotherapists working in the hospital. Knee functions will be evaluated with the IKDC scale, reaction time will be assessed with video recording supported by the Kinovea program, kinesiophobia will be assessed with the Tampa kinesiophobia scale, and finally, autonomic functions will be evaluated with the polar device. Measurements will be repeated after 6 weeks of interventions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with anterior cruciate ligament repair,
* Individuals who have no experience in this type of training,
* Not having any vision, hearing, or speech problems that would prevent the tests from being performed.
* Individuals who agree to the purposes of this study and to participate voluntarily.

Exclusion Criteria:

* Have previous experience in Motor Imagery techniques or training,
* Having any orthopedic problem that prevents walking,
* Having a history of neurological disease,
* People being treated with any medication that affects the central nervous system

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia | Through study completion, an average of 1 year
  Tampa Kinesiophobia Scale: This scale, consisting of 17 questions, evaluates the person's avoidance of movement or fear of re-injury. A Likert-type scale consisting of 4 points is used. 1 point means 'I disagree', and 4 points means 'I agree'. The individual receives a total score between 17 and 68 on this scale. A high score means high kinesiophobia.
Activity Level | Through study completion, an average of 1 year
  Tegner Activity Scale: Although the scale consists of 11 questions in total, the difficulty level increases as you go from 0 to 10. While 0 means that he is either resting or retired due to his knee problem, 10 means that he is at a level where he can play competitive football at the national and elite levels. The individual is asked to mark the most appropriate one among these 11 items according to his activity level.

SECONDARY OUTCOMES:
Knee Fuctions | Through study completion, an average of 1 year
  IKDC (International Knee Documentation Committee): The IKDC is a purely subjective assessment that assigns patients a functional overall rating. Three categories are examined by the questionnaire: symptoms, athletic activity, and knee function. The symptoms subscale aids in evaluating issues like pain, stiffness, edema, and knee giving way. The stair climbing, standing up from a chair, squatting, and jumping functions are the emphasis of the sports activity subscale. Higher scores indicate higher levels of function and lower levels of symptoms, with the transformed score being regarded as a measure of function.
Self-confidence Level | Through study completion, an average of 1 year
  Athletic Injury Self-Efficacy Questionnaire (AISEQ): The questionnaire comprised 10 items representing 3 types of self-efficacy: task (3 items), barrier (3 items), and scheduling (4 items). Participants rate their self-efficacy for each of the items on a confidence scale ranging from 0% (no confidence) to 100% (completely confident).

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Işıntaş, Study Director — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)